CLINICAL TRIAL: NCT05193734
Title: A Phase II/III Randomized, Double-blind Controlled Study to Compare the Safety and Immunogenicity of 1 or 2 Doses of Acellular Pertussis Vaccines Containing Genetically-detoxified Pertussis Toxin in Young Adults Previously Primed With Acellular Pertussis Vaccines
Brief Title: Safety and Immunogenicity of 2 Doses Versus 1 Dose of Acellular Pertussis Vaccines Containing Genetically-detoxified Pertussis Toxin in Young Adults Previously Primed With Acellular Pertussis Vaccines
Acronym: Pertagen2x
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Blanchard-Rohner Geraldine, Principal Investigator, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PERTAGEN2x
Record Dates: First submitted 2021-11-23; First posted 2022-01-18 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Pertussis; Vaccine-Preventable Diseases
MeSH Terms: conditions — Whooping Cough; Vaccine-Preventable Diseases | interventions — FHD

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Pertagen (Experimental)
  Interventions: Drug: Pertagen®
- Group Control (Active Comparator)
  Interventions: Drug: Revaxis®

INTERVENTIONS:
Drug: Pertagen® — Schedule:
  Group Pertagen will receive two doses of Pertagen®. (one vaccination on Day 0 and 6 months later for each volunteer.)
  Mode of Administration:
  Intramuscular injection into the deltoid region of the upper extremity, using a syringe with a 1 to 1.5 inch #25-gauge sterile needle.
  Other Names: Genetically detoxified pertussis toxin (rPT) and filamentous hemagglutinin (FHA), alum adsorbed
  Arms: Group Pertagen
Drug: Revaxis® — Schedule:
  Group Control will receive one dose of Revaxis® on Day 0 followed by 1 dose of Pertagen® 6 months later for each volunteer.
  Mode of Administration:
  Intramuscular injection into the deltoid region of the upper extremity, using a syringe with a 1 to 1.5 inch #25-gauge sterile needle.
  Arms: Group Control

SUMMARY:
A significant increase of pertussis incidence is reported in a growing number of countries. This resurgence is considered as resulting from the limited durability of aP-vaccine-induced immunity and is associated with increased mortality in young infants and morbidity at all age groups. As the pertussis immunity acquired through immunization or infection is short-lived, its maintenance or reactivation requires repeat boosting at regular time points. Thus, novel strategies capable of reactivating pertussis immunity are needed.

The efficacy of current acellular pertussis vaccines (which contain chemically-detoxified pertussis toxoid (PT)) rapidly wanes, in part because priming and repeat immunization with acellular vaccines induce antibodies specific for the chemically-detoxified PT but unable to efficiently recognize the native PT expressed by B. pertussis.

Clinical studies have shown the superior immunogenicity profile of acellular pertussis vaccines including genetically-detoxified PT (rPT) in adults and adolescents previously primed with aP. In particular, the investigators showed in a past Geneva study in teenagers previously primed with aP that rPT/FHA induced a stronger recall response than the current aP-vaccine at one month post-vaccination. However, the difference was less clear one year after vaccination, suggesting that 2 doses may be needed for more sustained immunity.

In the present study, the investigators would like to assess whether giving two doses of rPT/FHA at 6 months interval induces stronger immune responses than a single dose.

ELIGIBILITY:
Inclusion Criteria:

* Has provided written informed consent;
* Male or female, ages 18 to 30 years (inclusive) at the time of enrollment;
* With documented history of acellular pertussis immunization (5 doses);
* Free of clinically significant health problems, as determined by pertinent medical history and clinical examination at study screening;
* Non-pregnant, non-lactating females :
* Able to attend all scheduled visits during one year and to understand and comply with the study procedures;

Exclusion Criteria:

* Prior dTpa immunization within the last 5 years or prior dT immunization within the last 2 years, or any other investigational vaccine likely to impact on interpretation of the trial data
* Suspected or confirmed pertussis infection within the last 10 years or documented pertussis infection in a household member within the last 10 years;
* History of severe local or systemic reactions to any vaccination;
* Known hypersensitivity or allergy to diphtheria, tetanus, or pertussis-containing vaccines (including excipients);
* Receipt of investigational product up to 30 days prior to enrollment or ongoing participation in another interventional clinical trial;
* Receipt of licensed vaccines within 30 days of planned study immunization or ongoing participation in another clinical interventional trial likely to interfere with study results;
* Acute or chronic, clinically significant psychiatric, hematologic, pulmonary, cardiovascular, or hepatic or renal functional abnormality as determined by the Investigator based on medical history and physical exam;
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection, asplenia, cytotoxic therapy in the previous 5 years, and/or diabetes;
* Has a known history of vaccine-induced Guillain-Barré Syndrome;
* Has an active malignancy or recent (<10 years) history of metastatic or hematologic malignancy;
* Suspected or known alcohol and/or illicit drug abuse within the past 5 years;
* Pregnant or lactating female, or female intending to becoming pregnant during the study period;
* Administration of immunoglobulins within the 120 days preceding study entry or planned administration during the study period;
* History of blood donation (at least 450 ml) within 30 days of enrollment or plans to donate within the 30 days following and preceding each blood draw;
* Receipt of chronic (>14 days) immunosuppressants or other immune-modifying drugs within 6 months of study entry:
* Any other significant finding that, in the opinion of the investigator, would increase the risk of the individual's having an adverse outcome by participating in this study.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-02-07 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity of two doses compared to a single dose of an acellular pertussis vaccine | 1 year
  The primary objective is to assess the immunogenicity of two doses compared to a single dose of an acellular pertussis vaccine (Pertagen®) including genetically-detoxified pertussis toxin (rPT) administered at 6 months interval and delivered by the intramuscular route to adults aged 18-30 years previously primed and boosted with chemically-detoxified PT.
  The main immunogenicity endpoints will be the geometric mean concentration (GMC) of anti-PT neutralizing antibodies assessed 4 weeks (early immunity) and 6 months (sustained immunity) following one or two injections of Pertagen® given at 6 months interval

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events OBJECTIVE | Solicited local and systemic reactions will be followed up for 7 days and AEs for 28 days after vaccination
  Safety endpoints evaluated by solicited local and systemic reactions and unsolicited adverse events (AEs)
Humoral immune response | At 28 days after vaccination
  GMCs and seroresponse rates of PT, FHA, tetanus and diphtheria-toxoid specific IgG antibodies measured by ELISA and specific elicited by two doses of Pertagen® as compared to a single dose.
Cellular immune response | At 28 days after vaccination
  Concentration of specific memory B cells for PT, tetanus

CONTACTS AND LOCATIONS:
Overall Officials: BLANCHARD ROHNER Geraldine, MD, Principal Investigator — University of Geneva
Locations (1):
- University of Geneva, Geneva, Switzerland

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-23): https://cdn.clinicaltrials.gov/large-docs/34/NCT05193734/Prot_SAP_000.pdf